CLINICAL TRIAL: NCT02959333
Title: Human Amniotic Epithelial Cells for Treatment of Bronchial Fistula
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hAEC-BF
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Bronchial Fistula
MeSH Terms: conditions — Bronchial Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hAEC treatment (Experimental): hAEC: human amniotic epithelial cells 3-5*10^7 /5 ml
  Interventions: Biological: hAEC

INTERVENTIONS:
Biological: hAEC — hAEC: human amniotic epithelial cells

SUMMARY:
Bronchial fistula (BF), an abnormal passage or communication between a bronchus and another part of the body, may develop when there are penetrating wounds of the thorax and after lung surgery. Without effective therapy, treatment of BF is a challenge, with a high rate of mortality and teratogenicity.

The investigators will conduct endoscopic injection of human amniotic epithelial cells to fistula, observe the recovery of bronchial fistula and systemic reactions, to investigate the application of human amniotic epithelial cells in the treatment of bronchial fistula.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bronchial fistula by Imaging or bronchoscopic examination
* typical symptom of bronchial fistula, such as fever, cough, purulent sputum, weight loss…
* patients present compromised conditions, who can only accept a conservative treatment.

Exclusion Criteria:

* absolute contraindication of bronchoscopic examination and treatment
* with previous treatment of cell therapy, including stem cells.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
median time for fistula closure | 12 weeks

SECONDARY OUTCOMES:
complication | 1 year
  fever, coughing up blood, infection...

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Zeng, Dr., Principal Investigator — The Second Affiliated Hospital of Fujian Medical University
Locations (1):
- The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided